CLINICAL TRIAL: NCT06247124
Title: OPERATION WIPE OUT: Multi-Channel Communication Campaign to Promote HPV Vaccination in Chambers County, Alabama
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB3000011735; P30CA013148 (NIH)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HPV Vaccination
Keywords: HPV vaccination; Schools; High school students

STUDY DESIGN:
Intervention Model Description: high school students are enrolled as research participants to develop a multi-channel campaign to promote HPV vaccination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV vaccination (Other): Multi-channel campaign to promote HPV vaccination
  Interventions: Behavioral: multi-channel communication campaign to promote HPV vaccination

INTERVENTIONS:
Behavioral: multi-channel communication campaign to promote HPV vaccination — High school students will develop, implement, and evaluate a multi-channel communication campaign to promote HPV vaccination.

SUMMARY:
The Advisory Committee on Immunization Practices (ACIP) recommends HPV vaccination for all children and adults ages 9 to 26 in the U.S. However, HPV vaccination rates nationally and in Alabama lag far behind the Healthy People 2020 goal of 80% coverage. Despite multiple efforts, Alabama still ranks third in cervical cancer mortality and incidence nationally with great disparities within the state, particularly between urban and rural counties. In order to address this public health challenge, organizations have come together to develop, implement, and evaluate a statewide action plan to eliminate cervical cancer as a public health problem in Alabama by 2033. This plan was officially launched by the State Health Officer in May 2023 as a partnership between government, academia, civic organizations, and non-profit organizations and is known as OPERATION WIPE OUT. The overall goal of this Supplement is to develop, implement, and examine the feasibility and scalability of a theory-driven, participatory multi-channel communication campaign to promote HPV vaccination uptake that is designed and delivered by high school students with the support of OPERATION WIPE OUT partners and linked to school-based vaccination in a rural county that has the highest cervical cancer incidence in the state (Chambers County). The specific aims are: (1) To develop and examine the feasibility of a theory-driven, participatory multi-channel communication campaign to promote HPV vaccination uptake with high school students being agents of change and provision of school-based vaccination; and (2) To examine specific features of the multi-channel communication campaign regarding scalability, sustainability, and potentially a future full-scale implementation science trial. The primary outcome will be HPV vaccination uptake at the county level obtained Alabama Department of Public Health Vaccination Registry (ImmPRINT). Additionally, treatment fidelity and scalability assessments will be conducted to inform sustainability efforts.

DETAILED DESCRIPTION:
The human papillomavirus (HPV) is the most common sexually transmitted infection in the U.S., and it has been well established that high-risk HPV infection is causally related to cervical, vaginal, vulvar, anal, and oropharyngeal cancer. This discovery led to the development of a safe and effective preventive vaccine that is available in U.S. through most health insurances or federally-funded programs. The Advisory Committee on Immunization Practices (ACIP) recommends HPV vaccination for all children and adults ages 9 to 26 in the U.S. However, HPV vaccination rates nationally and in Alabama lag far behind the Healthy People 2020 goal of 80% coverage. Despite multiple efforts, Alabama still ranks third in cervical cancer mortality and incidence nationally with great disparities within the state, particularly between urban and rural counties. In order to address this public health challenge, organizations have come together to develop, implement, and evaluate a statewide action plan to eliminate cervical cancer as a public health problem in Alabama by 2033. This plan was officially launched by the State Health Officer in May 2023 as a partnership between government, academia, civic organizations, and non-profit organizations and is known as OPERATION WIPE OUT. While the plan is comprehensive and outlines specific evidence-based strategies to promote HPV vaccination along with cervical cancer screening/follow-up, the evidence on multi-channel communication interventions (besides provider-focused interventions) to promote HPV vaccination uptake at the population level is scarce, and the results are mixed. The overall goal of this Supplement is to develop, implement, and examine the feasibility and scalability of a theory-driven, participatory multi-channel communication campaign to promote HPV vaccination uptake that is designed and delivered by high school students with the support of OPERATION WIPE OUT partners and linked to school-based vaccination in a rural county that has the highest cervical cancer incidence in the state (Chambers County). Key components will include: (a) capacity building of high school students providing them with knowledge, skills, and support to develop and implement the campaign; (b) engagement of parents, teachers, school nurses, and school administrators); and (c) school-based vaccination. The specific aims are: (1) To develop and examine the feasibility of a theory-driven, participatory multi-channel communication campaign to promote HPV vaccination uptake with high school students being agents of change and provision of school-based vaccination; and (2) To examine specific features of the multi-channel communication campaign regarding scalability, sustainability, and potentially a future full-scale implementation science trial. The primary outcome will be HPV vaccination uptake at the county level. Alabama has a robust vaccination registry managed by Alabama Department of Public Health (ImmPRINT). Additionally, treatment fidelity and scalability assessments (acceptability, feasibility, potential reach and adoption, alignment with the strategic context) will be conducted to inform sustainability efforts.

ELIGIBILITY:
Inclusion Criteria:

* High school students enrolled in the Health Science Program at the Chambers County School District, Alabama

Exclusion Criteria:

-

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
HPV Vaccination at the county level | One year
  HPV vaccination uptake at the county level

SECONDARY OUTCOMES:
HPV vaccination at the school level | one year
  HPV vaccination at the school level

OTHER OUTCOMES:
Knowledge and confidence among the high school students | 6 months
  Pre- and post-training level of knowledge and confidence among the high school students participating in the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Scarinci, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Chambers County School District, Lafayette, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There are only have 29 students enrolled in the research. Thus, there is a need to keep confidentiality